CLINICAL TRIAL: NCT06275568
Title: Accelerating Healthcare Engagement in Healthy Food Interventions - Food Rx in High Risk Pregnant Mothers With About Fresh and Community Health Choice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Heart Association (Other); Michael and Susan Dell Foundation (Unknown); Tufts University (Other)
Responsible Party: Principal Investigator, Shreela V Sharma, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC-SPH-23-0655
Record Dates: First submitted 2023-11-03; First posted 2024-02-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Nutrition in High-Risk Pregnancy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care Fresh Connect cardholder engagement (Active Comparator)
  Interventions: Behavioral: Usual Care Fresh Connect cardholder engagement
- Usual care Fresh Connect cardholder engagement plus Enhanced engagement communication (Experimental)
  Interventions: Behavioral: Usual Care Fresh Connect cardholder engagement; Behavioral: Enhanced engagement communication

INTERVENTIONS:
Behavioral: Usual Care Fresh Connect cardholder engagement — Fresh Connect, a Food as Medicine product of the non-profit organization About Fresh, Inc., consists of a pre paid, programmable debit card, a cloud-based cardholder success platform, and an analytic engine designed to illuminate the healthcare value of improved food access and nutritional security.
  This arm receives:
  * About Fresh Food Rx debit card ($100 per month from enrollment until 2 months post-partum)
  * Texts for all cardholders per month (1-2 outbound texts)
  * Welcome call from About Fresh cardholder engagement team
  * 1 text - notification that Fresh Connect funds have been reloaded
  * As-needed program updates (e.g. new retailers), inactivity outreach
  * Additional texts that would be ad hocs: texts with food experiences (cooking videos), produce how-tos, and fun engagement; and satisfaction surveys - e.g. feedback on the Fresh Connect program, feedback on retailers, satisfaction with cardholder success, etc.
Behavioral: Enhanced engagement communication — Enhanced engagement involves additional outbound texts per month and additional ad hoc bi-monthly or quarterly texts, as well as tailored reminder text to use funds before the end of the month.
  Arms: Usual care Fresh Connect cardholder engagement plus Enhanced engagement communication

SUMMARY:
The purpose of the study is to assess if the Fresh Connect food prescription (Fresh Connect Food Rx) program that provides consistent access to healthy fresh produce through purchases at the grocery store plus nutrition education impacts gestational weight gain, other pregnancy and birth outcomes, and food and nutrition security in low-income, ethnically diverse, at-risk women residing in Houston, Texas. Enrollment of participants will begin in pregnancy at the time of the first prenatal visit (as long as the first visit occurs before the end of the first trimester); each participant will be followed until 60 days post-partum (up to 11 months follow-up per participant).

ELIGIBILITY:
Inclusion Criteria:

* high-risk pregnant mothers receiving care at Texas Children's Health Plan (TCHP) managed care organizations in Houston, Texas
* <20 weeks medically confirmed viable pregnancy
* overweight/obese pre-pregnancy or at first trimester (self-report or measured BMI>30.0), and/or prior history of diabetes or gestational diabetes, and/or prior history of hypertension or pregnancy-induced hypertension

Exclusion Criteria:

* not a high-risk pregnant mother receiving care at Texas Children's Health Plan (TCHP) managed care organizations in Houston, Texas

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 620 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Absolute gestational weight gain (GWG) in pounds | From the start of the first trimester of pregnancy to the end of the first trimester of pregnancy (3 months)
Absolute gestational weight gain (GWG) in pounds | From the start of the second trimester of pregnancy to the end of the second trimester of pregnancy (3 months)
Absolute gestational weight gain (GWG) in pounds | From the start of the third trimester of pregnancy to the end of the third trimester of pregnancy (3 months)
Excess gestational weight gain (EGWG) in pounds | From the start of the first trimester of pregnancy to the end of the first trimester of pregnancy (3 months)
Excess gestational weight gain (EGWG) in pounds | From the start of the second trimester of pregnancy to the end of the second trimester of pregnancy (3 months)
Excess gestational weight gain (EGWG) in pounds | From the start of the third trimester of pregnancy to the end of the third trimester of pregnancy (3 months)

SECONDARY OUTCOMES:
Number of participants diagnosed with pregnancy-induced hypertension | From the time of enrollment until the time of birth (up to 9 months)
Number of participants diagnosed with gestational diabetes | From the time of enrollment until the time of birth (up to 9 months)
Number of participants with pre-term birth (<37 weeks) | at the time of birth
Infant birth weight | at the time of birth

CONTACTS AND LOCATIONS:
Overall Officials: Shreela Sharma, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
At the end of the project, de-identified data at individual level will be uploaded to the American Heart Association (AHA) Precision-Medicine Platform.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: June 2025
Access Criteria: Will be determined by AHA.

REFERENCES:
- See also: about Fresh Connect — https://www.aboutfresh.org/fresh-connect/